CLINICAL TRIAL: NCT06298240
Title: The Implementation of Nurse Demand Management as a Factor in Improving the Quality of Care in a Primary Care Emergency Center.
Brief Title: Implementation of Nursing Demand Management as a Factor for Improvement in a Primary Care Emergency Center.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4R22/074
Record Dates: First submitted 2024-02-06; First posted 2024-03-07 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-02

CONDITIONS: Nurse's Role; Disease, Acute
Keywords: primary care nursing; primary health care; nurses; acute disease/nursing; advanced rractice nursing; minor health problems; practice guideline
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consensuated nurse intervencion group (Experimental): Application of a consensual nursing guide with 5 reasons for health consultation where an autonomous role can be applied. Users who come to the emergency center during the first fifteen days of each month are assigned to the experimental group until the necessary sample of 156 subjects is reached.
  Interventions: Other: nursing procedure for acute health problems of low complexity
- Usual medical visit group (No Intervention): Users who come to the emergency center in the second fortnight of each month are assigned to the non-intervention (control) group where the usual medical visit is applied until the required sample of 156 subjects is reached.

INTERVENTIONS:
Other: nursing procedure for acute health problems of low complexity — An agreed nursing procedure is applied for users of a primary care emergency center who spontaneously consult for 5 acute health problems of low complexity: gastroenteritis, cystitis in women, dental pain, upper respiratory tract affections and acute wounds
  Arms: Consensuated nurse intervencion group

SUMMARY:
Background: Nurse Demand Management was born in 2009 out of the need to address the growth of spontaneous acute demand in primary care. But it is not until 2013 that guidelines for the exercise of nursing actions in demand management were established in Catalonia, Spain. Nurses trained specifically to solve acute and low complexity health problems generate a quality of care comparable to that provided by family medicine doctors. On the other hand, it is worth highlighting the need to rationalise medical resources in primary care centres, primary care emergency centres or points of continuous care (different emergency facilities in the territory in terms of size and services) in order to give priority to doctors being able to dedicate more time to medium or high complexity pathology. Although nurse demand management has been implemented in primary care teams for years, it is being carried out in different intensities according to the needs or priorities of each health territory.

The promotion of the autonomous role of nursing through the implementation of nurse demand management in the urgent spontaneous demand of low complexity can be transcendent, both in the optimisation of health resources in primary care and in the management of the demand for care.

Hypothesis: The implementation of nurse demand management is a factor of improvement in the efficiency and quality of care in the Primary Care Emergency Centre of the city of Mataró (Barcelona, Spain). Objectives: The main objective of this study was to determine whether the implementation of nurse demand management is a factor in improving efficiency and quality of care in the CUAP of Mataró. Methodology: Non-randomised controlled experimental intervention study. Application of a consensual guide with 5 reasons for health consultations where demand management nursing can be applied.

DETAILED DESCRIPTION:
Background: Demand Nurse Management was born in 2009 due to the need to address the growth of spontaneous acute demand in primary care. But it was not until 2013 that guidelines for the practice of demand management nursing were established in Catalonia, Spain. Nurses trained specifically to solve acute and low complexity health problems generate a quality of care comparable to that provided by family medicine physicians. On the other hand, it is worth highlighting the need to rationalize medical resources in primary care centers, primary care emergency centers or points of continuous care (different emergency devices in the territory in terms of size and services) in order to prioritize physicians' time for medium or high complexity pathology. Although nurse demand management has been implemented in primary care teams for years, it is being carried out in different intensities according to the needs or priorities of each health territory. The most complete research work, to date, regarding demand management nursing, was carried out between 2011 and 2012 at the Can Bou primary care center in Castelldefels, Barcelona. A retrospective, observational, descriptive and cross-sectional study was conducted, which concluded that the application of demand management nursing showed a high resolution of diseases attended and a high percentage of health advice and health education in visits attended autonomously by nurses. Primary care emergency points and centers form a powerful network in the spontaneous urgent demand of low and medium complexity and help to stop the collapse of hospital care and make it easier for hospital care to focus on highly complex or vital emergencies. The promotion of the autonomous role of nursing through the implementation of nurse demand management in urgent spontaneous demand of low complexity can be transcendent, both in the optimization of health resources in primary care throughout the territory, as well as in the improvement in terms of the quality and efficiency of these services and the quality of care for their users. Hypothesis: The implementation of nurse demand management is a factor of improvement in the efficiency and quality of care in the Primary Care Emergency Center of the city of Mataró (Barcelona, Spain). Objectives: The main objective was to determine whether the implementation of demand management nursing is a factor for improving efficiency and quality of care in the CUAP of Mataró, and specifically, to evaluate whether it frees time for physicians to attend medium and high complexity health problems, reduces consultations for health problems attended within 15 days, the level of user satisfaction, and whether it facilitates efficiency and quality with respect to waiting time and resolution of the health problem. Methodology: Non-randomized controlled experimental intervention study. Application of a consensual guide with 5 health consultation reasons where the nursing management of the demand can be applied the first fifteen days of each month in the emergency center of Mataró (experimental group) and until reaching the necessary sample of 156 subjects. Control group of application in the second fortnight of each more where the usual operation is applied and until reaching a necessary sample of 156 subjects. Determinations: Sociodemographic, clinical data, characteristics of the visits and patient experience will be collected. Statistical analysis: Descriptive, correlational and multivariate analysis will be performed. Expected results: Improvement in waiting time, resolution, number of consultations and user satisfaction with respect to low intensity health consultations under the application of nurse demand management. Improved efficiency of the emergency center and quality of care of the service. Applicability and Relevance: This is a first prospective experimental study that may help public health authorities to determine the general interest in the widespread implementation of demand management nursing in emergency and non-emergency primary care.

ELIGIBILITY:
Inclusion Criteria:

* All users who come to the emergency centre between Monday and Friday (excluding public holidays) from 8 a.m. to 8 p.m. and who consult for the 5 possible health problems that are part of the study protocol.

Exclusion Criteria:

* Any spontaneous user or user referred by another health centre who comes for a re-consultation for the same health problem in less than 30 days will be excluded.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Waiting time and resolution of the visit | During the entire process of assistance to the participant, an average of 4 hours.
  Different time points are collected to analyze the duration of care at the center: time of entry into the triage consultation, time of entry into the medical or nursing consultation, and time of departure from the consultation.
  Time that the administrator receives the user and includes him/her in the work agenda of the emergency center.
  Time the user makes the triage. Time that the user is attended in the agenda of the demand management center (experimental group days).
  Time that the user is seen in the medical office (control group days).
Number of reconsultations | 30 days
  Number of return visits for the same health problem made by the participant in the subsequent 30 days.
patient experience | On a scale from 0 to 10, where 0 is not very satisfied and 10 is very satisfied.
  Participant satisfaction survey, on the same day, of the care received by the doctor or nurse From 15 days after the hearing, a quality telephone survey will be conducted with all recruited subjects.

OTHER OUTCOMES:
Prescribed drugs | 0 to 10
  number of drugs
Processed labour disabilities | 0 to 1
  Number of processed labour disabilities
Diagnoses change | 0 to 1
  Diagnoses change at the visits for the same health problem fort the next month

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Estarlich Corominas, IP, Principal Investigator — Active nurse in the emergency center where the study is carried out
Locations (1):
- Mataró primary care emergency center, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estarlich-Corominas J, Soler-Abril N, Casanellas-Chuecos A, Becerra-Corzo S, Bianco AS, Toran-Monserrat P, Garcia-Sierra R. Nurse management of minor problems in primary care emergencies: a non-randomized controlled trial. BMC Nurs. 2025 Jan 24;24(1):87. doi: 10.1186/s12912-025-02729-2. PMID 39856650